CLINICAL TRIAL: NCT03768440
Title: Continuous Erector Spinae Block Versus Continuous Paravertebral Block Following Thoracotomy: A Randomized, Controlled Non-Inferiority Study
Brief Title: Continuous Erector Spinae Block Versus Continuous Paravertebral Block
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: LACK OF INTEREST
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Roland Brusseau, Associate in Perioperative Anesthesia, Department of Anesthesiology, Perioperative and Pain Medicine Instructor in Anaesthesia, Havard Medical School, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB-P00030317
Record Dates: First submitted 2018-11-16; First posted 2018-12-07 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Pain, Postoperative
Keywords: ropivacaine infusion; regional anesthesia; paravertebral block; erector spinae block
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine; PVB protocol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- continuous erector spinae block (Experimental): An erector spinae block is placed at end of the thoracotomy procedure, bolused with 1ml/kg 0.2% ropivacaine, then started on a 0.2ml/kg/hour continuous infusion of 0.2% ropivacaine. patients will have access to rescue opiates as needed by means of the standard PCA/NCA demand protocols utilized at BCH. Rescue analgesic consumption will be tabulated at 24, 48 and 72 hours, rendered as total opiate equivalents.
  Interventions: Procedure: continuous erector spinae block (ESB); Drug: Ropivacaine
- continuous paravertebral block (Active Comparator): A paravertebral block is placed at end of the thoracotomy procedure, bolused with 1ml/kg 0.2% ropivacaine, then started on a 0.2ml/kg/hour continuous infusion of 0.2% ropivacaine. patients will have access to rescue opiates as needed by means of the standard PCA/NCA demand protocols utilized at BCH. Rescue analgesic consumption will be tabulated at 24, 48 and 72 hours, rendered as total opiate equivalents.
  Interventions: Procedure: continuous paravertebral block (PVB); Drug: Ropivacaine

INTERVENTIONS:
Procedure: continuous erector spinae block (ESB) — Erector spinae block: T4/5 transverse process is identified with the ultrasound transducer in a parasagittal orientation; the needle tip is advanced until it contacts the transverse process, just below the erector spinae muscle complex; the erector spinae muscle is visualized to be elevated up off of the transverse process with normal saline injection. Following a bolus injection of 2ml/kg of 0.2% ropivacaine, a catheter is threaded into the space occupied by the local anesthetic bolus.
  Other Names: ESB with ropivacaine; Naropin
  Arms: continuous erector spinae block
Procedure: continuous paravertebral block (PVB) — The paravertebral space (bound medially by the bodies of the vertebrae, intervertebral discs, and intervertebral foraminae; anterolaterally by the parietal pleura and the innermost intercostal membrane; posteriorly by the transverse processes of the thoracic vertebrae, heads of the ribs, and the superior costotransverse ligament) laying between T4/5 is identified using the ultrasound transducer in a transverse orientation; the needle tip is advanced until it is seen passing under the transverse process, immediately superior to the pleura; the pleura is seen to deflect downward with normal saline injection. Following a bolus injection of 2ml/kg of 0.2% ropivacaine, a catheter is threaded into the space occupied by the local anesthetic bolus.
  Other Names: PVB with ropivacaine; Naropin
  Arms: continuous paravertebral block
Drug: Ropivacaine — Ropivacaine 0.2% will be the drug used for each group (ESB group and PVB group)
  Other Names: Naropin

SUMMARY:
Overall Aim: To evaluate the efficacy of continuous erector spinae block (ESB) versus continuous paravertebral block (PVB) for postoperative analgesia in children and adolescents undergoing surgical procedures via unilateral thoracotomy.

Hypothesis: The investigators hypothesize that ESP block efficacy is not inferior to that of PVB with respect to pain control and consumed opiate equivalents at 24 hours postoperatively.

DETAILED DESCRIPTION:
Regional anesthesia-and pediatric regional anesthesia in particular-is a rapidly evolving subfield of anesthesia practice driven with considerable urgency by the growing recognition that even appropriate perioperative narcotic administration can have significant derogatory long-term effects.

Regional anesthetics can provide targeted, continuous analgesia to select dermatomes with minimal additional patient risk and have become routine components of opioid-sparing intraoperative and postoperative pain management plans for surgical patients at BCH. In addition to the postulated benefit of reducing overall opioid exposure and potentially reducing the risk for long term physiologic and behavioral dependence upon opioids, regional anesthetics may allow for earlier extubation after selected surgeries, shorter ICU, PACU and inpatient admissions, earlier mobilization, fewer gastrointestinal complications, and improved patient satisfaction scores.

Given the rapid evolution of the field of regional anesthesia and the fact that there are often multiple approaches for achieving analgesia in a select set of dermatomes, there are often a variety of regional anesthetic options for any given surgery. Some approaches are longstanding and well-studied, but with increasing frequency since the advent of ultrasound guidance, newer, novel nerve block options exist. As it is often expensive and work-intensive to thoroughly evaluate a given regional technique with a controlled pediatric trial, many of these blocks become standards of practice based on anecdote, retrospective analysis, or simply belief in the putative benefits of regional anesthetics.

The investigators are fortunate at BCH to have one of the largest concentrated pediatric surgical populations in the US. They also have an active, and well organized regional anesthesia service. Because of this, the investigators are in a unique position to more thoroughly evaluate the effectiveness and safety of regional anesthesia in children. Furthermore, the investigators feel it is critical that institutions such as BCH take a leading role in documenting the effects of regional anesthesia on the most important outcome measures when considering perioperative medicine. These include overall pain management, surgical healing, functional recovery, long-term pain symptoms, and emotional/behavioral outcomes after surgery.

Recently the ESB has become popular for providing analgesia after a number of anterior chest and abdominal procedures. This is a simple interfascial plane block that can reliably provide unilateral chest and/or abdominal wall analgesia. It has been described in numerous case reports and one case series as an effective block for management of unilateral thoracotomies, unilateral rib fractures, unilateral abdominal incisions and (when used bilaterally) for management of post-sternotomy pain.

As an interfascial plane block in a compressible anatomical space, the ESB is thought to be safe in anticoagulated (or recently anticoagulated) patients. It is fast becoming a preferred anesthetic option for these patients as opposed to neuraxial (e.g. epidural) and paraneuraxial (i.e. paravertebral) nerve blocks.

Given the ESB's potentially favorable risk profile versus the other blocks (it is technically less challenging, more distant from critical structures, and thought to be safe in anticoagulated patients) it could provide both a safer and easier to perform regional anesthesia option for many patients. It also offers a new option for a subset of anticoagulated patients for whom other regional techniques (epidural, paravertebral) are contraindicated.

Indeed, given the current information available related to the ESB, the regional anesthesia service at BCH has begun employing it when possible in circumstances where a PVB would commonly be used but is relatively or absolutely contraindicated. Patients undergoing thoracotomies while anticoagulated for cardiopulmonary bypass, aortic clamping, etc. have been successfully managed with continuous ESBs. In addition, thoracotomies in patients with acquired (e.g. dilutional) and other pathologic coagulopathies have been managed with ESBs. As such, the ESB has been adopted for routine use in specific patient populations at BCH and has even occasionally been utilized in lieu of the more longstanding routine PVBs or epidural blocks for patients without contraindication for such.

Retrospective review of BCH outcomes data for 47 ESBs done for a variety of surgeries and populations has not revealed any significant differences between PVBs and ESBs in terms of adverse events, postoperative opiate use, median pain scores, or other standard outcomes measures. As this data is observational in nature, it is difficult to draw firm conclusions as to the comparative efficacy of the two blocks. However, since there are differences in technical difficulty, relative contraindications, and there exist populations that might benefit from these blocks, it would be prudent to comparatively evaluate these blocks in a controlled, randomized, trial.

The investigators propose to evaluate the comparative efficacy of ESBs and PVBs for patients undergoing unilateral non-cardiac thoracotomy by means of a randomized, controlled non-inferiority study (based on a threshold of clinical significance being defined as a 15% difference) comparing rescue analgesic requirements, rendered as opiate equivalents, at 24 postoperatively. Rescue opiates will be available as needed by means of standard PCA/NCA demand protocols. Secondary measures will include rescue opiate requirements at 48 and 72 hours, pain scores, adverse events, time to discharge from the ICU, time to extubation, patient disposition after surgery, and time to perform the block in the operating room.

ELIGIBILITY:
Inclusion Criteria:

* ASA I - III status, undergoing unilateral thoracotomy for either esophageal atresia related intrathoracic procedures or other non-cardiac general surgical intrathoracic procedures.

Exclusion Criteria:

* Patients undergoing procedures including pleurodesis, pleural stripping, and decortication or other procedures with widely distributed pleural disruption.
* Patients with severe neurodevelopmental delays.
* Patients with previous chronic pain syndromes.
* Patients with a history of opioid treatment at any point in the 2 months prior to surgery.
* Lack of parental consent and/or child assent.

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2019-04-16 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Rescue analgesic consumption | 24 hours
  rescue opiates (rendered as morphine equivalents/kg) given by blinded providers using standard PCA/NCA demand protocols

SECONDARY OUTCOMES:
Pain scores | 24, 48 and 72 hours
  Pain scores measured by the numeric rating scale (NRS: 0/none -> 10/worst)
Time to perform the block in the operating room | 1 hour
  Total time required for intervention
Number of Adverse events | 1 week
  Any intervention related (or unrelated) adverse events
Rescue analgesic consumption | 48 hours
  rescue opiates (rendered as morphine equivalents/kg) given by blinded providers using standard PCA/NCA demand protocols
Rescue analgesic consumption | 72 hours
  rescue opiates (rendered as morphine equivalents/kg) given by blinded providers using standard PCA/NCA demand protocols

CONTACTS AND LOCATIONS:
Overall Officials: ROLAND BRUSSEAU, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children"S Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No